CLINICAL TRIAL: NCT01972269
Title: Determination of the Effective Volume of the 0.125% Bupivacaine-fentanyl 5mcg/mL Mixture Used for Epidural Analgesia in Labor
Brief Title: Determination of the Effective Volume of 0.125% Bupivacaine-fentanyl 5mcg/mL in Labour Epidurals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-06; 13-0247-A (Other: Research Ethics Board)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: Epidural; Labor Analgesia; Bupivacaine; Minimum effective volume
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (14):
- bupivacaine-fentanyl 4 (Active Comparator): Test dose: 3mL of 0.125% bupivacaine-fentanyl 5mcg/mL. Loading dose: 4mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl
- bupivacaine-fentanyl 6 (Active Comparator): Test dose: 3mL of 0.125% bupivacaine-fentanyl 5mcg/mL. Loading dose: 6mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl
- bupivacaine-fentanyl 8 (Active Comparator): Test dose: 3mL of 0.125% bupivacaine-fentanyl 5mcg/mL. Loading dose: 8mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl
- bupivacaine-fentanyl 10 (Active Comparator): Test dose: 3mL of 0.125% bupivacaine-fentanyl 5mcg/mL. Loading dose: 10mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl
- bupivacaine-fentanyl 12 (Active Comparator): Test dose: 3mL of 0.125% bupivacaine-fentanyl 5mcg/mL. Loading dose: 12mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl
- bupivacaine-fentanyl 14 (Active Comparator): Test dose: 3mL of 0.125% bupivacaine-fentanyl 5mcg/mL. Loading dose: 14mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl
- bupivacaine-fentanyl 16 (Active Comparator): Test dose: 3mL of 0.125% bupivacaine-fentanyl 5mcg/mL. Loading dose: 16mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl
- lidocaine 4 (Active Comparator): Test dose: 3mL of 2% lidocaine. Loading dose: 4mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl; Drug: Lidocaine
- lidocaine 6 (Active Comparator): Test dose: 3mL of 2% lidocaine. Loading dose: 6mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl; Drug: Lidocaine
- lidocaine 8 (Active Comparator): Test dose: 3mL of 2% lidocaine. Loading dose: 8mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl; Drug: Lidocaine
- lidocaine 10 (Active Comparator): Test dose: 3mL of 2% lidocaine. Loading dose: 10mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl; Drug: Lidocaine
- lidocaine 12 (Active Comparator): Test dose: 3mL of 2% lidocaine. Loading dose: 12mL of 0.125% bupivacaine-fentanyl 5mcg/mL.
  Interventions: Drug: Bupivacaine-fentanyl; Drug: Lidocaine
- lidocaine 14 (Active Comparator): Test dose: 3mL of 2% lidocaine. Loading dose: 14mL of 0.125% bupivacaine-fentanyl 5mcg/mL
  Interventions: Drug: Bupivacaine-fentanyl; Drug: Lidocaine
- lidocaine 16 (Active Comparator): Test dose: 3mL of 2% lidocaine. Loading dose: 16mL of 0.125% bupivacaine-fentanyl 5mcg/mL
  Interventions: Drug: Bupivacaine-fentanyl; Drug: Lidocaine

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — 0.125% bupivacaine-fentanyl 5mcg/mL
  Other Names: Marcaine
Drug: Lidocaine — 2% lidocaine
  Arms: lidocaine 10; lidocaine 12; lidocaine 14; lidocaine 16; lidocaine 4; lidocaine 6; lidocaine 8

SUMMARY:
Different medications can be used as analgesics in labor epidurals. Bupivacaine is one of the most commonly used drugs for that purpose. The efficacy of a certain medication injected epidurally depends on the dose that is given. A certain dose can be administered in different concentrations, which will consequently mean different volumes. Studies have been done to determine volumes for different concentrations of bupivacaine. However, those studies fall short in the sense that this information cannot be readily applicable in clinical practice, as we don't use bupivacaine plain. The combination of bupivacaine and fentanyl or sufentanil is common practice, as it is well established that the opioids will reduce the concentration of local anesthetic required to produce optimal effect with the least side effects.

This study is being planned to determine and compare the EV90 of the bupivacaine 0.125%-fentanyl mixture for initiation of labor epidural analgesia, following the administration of the 2 different test doses (3cc of lidocaine 2% or 3cc of the bupivacaine 0.125%-fentanyl mixture) used in our Department.

DETAILED DESCRIPTION:
Epidural administration of local anesthetics during labor produces analgesia, sympathetic block and motor block. The characteristics of the block depend on the volume and concentration of the local anesthetic that is used as well as the use of adjuncts(in our case: Fentanyl). Although many researchers have investigated the efficacy of different drugs at different concentrations, the volumes used have been arbitrary. There is limited data regarding the minimum volume that is necessary for a successful anesthetic for a given concentration of bupivacaine.

This study is conducted as a prospective, randomized, up-down sequential allocation trial. The aim is to determine the minimum volume of 0.125% bupivacaine in combination with 5mcgr/ml fentanyl that will provide effective analgesia for 90% of parturients in the first stage of labor. The verbal numeric rating scale (VNRS) is used to rate the pain felt over the first 20 minutes, where 0 is no pain and 10 is the worst pain imaginable. After 20 minutes, if the VNRS was greater than 1, the volume of the bupivacaine/fentanyl mixture was considered inadequate and additional volume of the mixture will be given.

After the randomised test dose of either 3cc lidocaine 2% or 3cc of the bupivacaine/fentanyl mixture is given, the loading volume of the bupivacaine/fentanyl mixture will be given. The volume of the bupivacaine/fentanyl mixture for the first patient was chosen at 10 ml (This is the volume with which is generally started in standard practice), and the dose for each subsequent patient depends on the outcome of the previous injection. Doses will be increased or decreased in increments of 2 ml. If the previous response was ineffective, the next patient will receive 2 ml more than the last patient. If the response of the previous patient is effective, the biased coin up-and-down allocation design, which is used to cluster doses around EV90, will be applied to determine if the dose remains the same or decreases.

40 patients will be included in each group within the study. The target volume, EV90, which is defined as the volume at which adequate response would occur in 90% of patients, will be estimated for each of the two test dose groups using Dixon and Mood method. The 95% confidence interval of EV90s will be estimated and based in comparing the EV90 between two groups. Isotonic Regression method will also be conducted to assess the EV90s. The side effects will also be summarized by the volume levels descriptively.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Full term (minimum 37 weeks gestation)
* Singleton pregnancy, vertex presentation
* Regular painful contractions occurring at least every 5 minutes
* VAS Pain score at requesting analgesia > 5 (VNPS 0-10)
* Cervical dilatation < 5 cm

Exclusion Criteria:

* Refusal to provide written informed consent.
* Any contraindication to epidural anesthesia
* Accidental dural puncture
* Allergy or hypersensitivity to bupivacaine or fentanyl
* Use of opioids or sedatives within the last 4 hours.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
VNRS pain score | 20 minutes
  The efficacy of the loading dose will be defined as a pain score ≤ 1 at 20 minutes following injection of the loading dose.

SECONDARY OUTCOMES:
Dermatome sensory level | 20 min
  Dermatome sensory level measured using ice
Motor block | 20 min
  Measured by modified Bromage score; 0 = no impairment, 1 = unable to raise the extended leg but able to move/flex knees and feet, 2 = unable to raise extended leg or flex knees, but able to move foot, 3 = unable to flex ankle, feet or knees).
Hypotension | 20 min
  Hypotension, defined as a drop in systolic blood pressure greater than 20% from baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada